CLINICAL TRIAL: NCT05398614
Title: Early Clinical Study of SENL101 Autologous T Cell Injection in the Treatment of Adult Patients With Relapsed or Refractory CD7+ Hematolymphoid Malignancies
Brief Title: SENL101 Autologous T Cell Injection in Adults With Relapsed or Refractory CD7+ Hematolymphoid Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SENL101 for CD7+
Record Dates: First submitted 2022-05-20; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: T-ALL; Lymphoma, T-Cell
Keywords: CD7; T-ALL/T-LBL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T (Experimental): SENL101
  Interventions: Biological: SENL101

INTERVENTIONS:
Biological: SENL101 — Patients will be treated with CD7 CAR-T cells

SUMMARY:
To evaluate the tolerability and safety of SENL101 in patients with relapsed or refractory CD7+ hematolymphoid malignancies.

DETAILED DESCRIPTION:
Main research purposes:

To evaluate the tolerability and safety of SENL101 in patients with relapsed or refractory CD7+ hematolymphoid malignancies.

Secondary research purposes:

To preliminarily evaluate the efficacy, pharmacokinetics and pharmacodynamics of SENL101 in the treatment of patients with relapsed or refractory CD7+ hemolymphoid malignancies.

Exploratory research purpose：

1. To explore the immunogenicity of SENL101；
2. T cell NK cell recovery time after treatment；
3. Other indicators of interest to researchers。

ELIGIBILITY:
The subjects of this study were patients with recurrent or refractory hematocratic malignancies of CD7+.

Inclusion Criteria:

1. Subjects diagnosed with refractory/relapsing T-cell leukaemia/lymphoma met one of the following criteria: relapse: disease recurrence after complete remission with at least two prior regiments or complete remission with stem cell transplantation; Refractory: patients who have received at least two previous treatment regimens and failed to achieve a complete or partial response after the last treatment (leukemia patients), or failed to achieve a response after stem cell transplantation or develop disease progression;
2. The tumor cells detected by bone marrow flow cytometry were CD7+ and/or extramedullary lesions were diagnosed as CD7+ by pathological immunohistochemistry at the time of enrollment and screening;
3. If tumor cells were detected in peripheral blood during enrollment and screening, it was required to meet the requirement that the surface immunophenotype of tumor cells was CD4 and CD8 double negative by flow cytometry. If the surface phenotype of peripheral blood tumor cells was not CD4 and CD8 double negative, the proportion of tumor cells in peripheral blood was ≤1%;
4. Life expectancy greater than 12 weeks;
5. ECOG 0-2;
6. Age 18-65 (upper and lower limits included);
7. HGB at least 70g/L,PLT 20x109/L, can be transfused;
8. Liver and kidney functions The cardiopulmonary functions meet the following requirements: Oxygen saturation under air ≥ 92%; LVEF≥45%; Total bilirubin <3×ULN; ALT/AST<5×ULN; Creatinine <1.5×ULN;
9. Informed consent explained to, understood by and signed by patient/ guardian.

Exclusion Criteria:

Those who meet any of the following criteria are not eligible to join the group:

1. New York Heart Association (NYHA) classification ≥ grade III heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris or other clinically prominent heart disease within one year before signing the informed consent form, Or QTc interval >480ms at screening (QTc interval calculated by Fridericia formula);
2. If the patient has a history of hematopoietic stem cell transplantation, 6 months after the patient received allogeneic hematopoietic stem cell transplantation;
3. Those with active GvHD or those who require immunosuppressive therapy;
4. Malignancy other than T-cell acute lymphoblastic leukemia/lymphoma within 5 years prior to screening, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer after radical surgery, radical surgery ductal carcinoma in situ;
5. Active or uncontrollable infection requiring systemic treatment within 7 days prior to screening (except for mild urogenital infections and upper respiratory tract infections);
6. History of autoimmune disease (eg, rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease) requiring systemic immunosuppressive/systemic disease modulating medication within the past 2 years;
7. When screening, if the hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HbcAb) is positive, and the peripheral blood hepatitis B virus (HBV) DNA is higher than the detection limit, it needs to be excluded; if the hepatitis C virus (HCV) antibody is positive, the peripheral blood HCV Those with positive RNA need to be excluded; those with positive human immunodeficiency virus (HIV) antibody; those with positive cytomegalovirus (CMV) DNA test; those with positive test for Treponema pallidum specific antibody (TPPA) need to be excluded;
8. Participate in other clinical trials within 4 weeks before the informed consent is signed, or the date of the informed consent is signed and the last medication of the drug is still within 5 half-lives of the drug (whichever is longer);
9. History of severe allergy to biological products;
10. Unstable systemic disease as judged by the investigator: including but not limited to severe liver, kidney or metabolic disease requiring drug therapy;
11. Pregnant or breastfeeding women, and female subjects planning pregnancy within 2 years of cell infusion or male subjects whose partner is planning pregnancy within 2 years of cell infusion;
12. Subjects who have received CAR-T therapy or other gene-modified cell therapy prior to screening;
13. Circumstances that the investigator believes may increase the risk to the subject or interfere with the results of the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | 24 months post CAR-T cells infusion
  The incidence and severity of adverse events and adverse reactions from infusion to withdrawal or before the safety follow-up period

OTHER OUTCOMES:
Cytokine release | 12 months post CAR-T cells infusion
  Changes from baseline in IFN-γ, TNF-α, IL-2, IL-6, IL-10
CD7 positive cells in peripheral blood at each time point | 12 months post CAR-T cells infusion
  Absolute value and ratio of CD7 positive cells (T cells NK cells) at each time point in peripheral blood
T cell subsets | 12 months post CAR-T cells infusion
  T cell subsets monitoring at each time point (CD4+ CD8+ CD4+/ CD8+ ratio)
Immunogenicity endpoint | 12 months post CAR-T cells infusion
  Detectable antibody concentration in serum at each time point
T cell NK cell recovery time after treatment | 12 months post CAR-T cells infusion
  Absolute value of T cells NK cells at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Liang Huang, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China